CLINICAL TRIAL: NCT05603078
Title: A Prospective Study of Preoperative MRI Linac-based Tumor-bed Boost Followed by Breast-conservative Oncoplastic Surgery and Adjuvant Ultra-hypofractionated Whole Breast Radiotherapy for Early Stage Breast Cancer
Brief Title: A Prospective Study of Preoperative Tumor-bed Boost Followed by Oncoplastic Surgery and Adjuvant Whole Breast Radiotherapy for Early Stage Breast Cancer (BIRKIN)
Acronym: BIRKIN
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other)
Responsible Party: Principal Investigator, HAO JING, professor of medicine, Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCC2021291
Record Dates: First submitted 2022-10-22; First posted 2022-11-02 (Actual); Last update posted 2022-11-02 (Actual); Status verified 2022-10

CONDITIONS: Breast Neoplasms
Keywords: Breast cancer; MRI guided radiotherapy; Pre-operative radiotherapy; Ultra-hypofractionation
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- preoperative tumor-bed boost (Experimental): The participants receive preoperative tumor-bed boost, oncoplastic surgery and adjuvant WBRT±RNI.
  Interventions: Radiation: Preoperative MRI-guided tumor-bed boost and postopreative ultra-hypofractionated radiotherapy (26 Gy/5.2Gy/5)

INTERVENTIONS:
Radiation: Preoperative MRI-guided tumor-bed boost and postopreative ultra-hypofractionated radiotherapy (26 Gy/5.2Gy/5) — Preoperative tumor-bed boost was performed under MRI Linac, and a single dose of 10Gy is prescribed. The postoperative radiotherapy of 26Gy/5.2Gy/5 fractions is within 6 weeks following surgery. Adjuvant chemotherapy, targeted therapy and endocrine therapy are initiated no more than 12 weeks after surgery.

SUMMARY:
This study explores the feasibility of preoperative single-dose tumor-bed boost followed by oncoplastic breast-conserving surgery and ultra-hypofractionated postoperative radiotherapy in patients with early stage breast cancer. Patients less than 55 years old, who are diagnosed with breast cancer and are eligible to recieve breast-conserving surgery are enrolled. Patients who are older than 55 years, with suspected regional lymph node metastasis are excluded. The primary end point are the acute toxicities within 4 weeks after adjuvant radiation. The secondary endpoints are oncologic outcomes, surgical complications within 30 days, late toxicities, patients' quality of life and cosmetic outcomes.

DETAILED DESCRIPTION:
This is a prospective, non-controlled, feasitility study. The tumor-bed boost part of the radiotherpay is put forward, 7-14 days before the definitive surgery. A single dose of 10Gy is prescribed to the tumor bed. In order to identify the tumor accurately, MRI guided radiotherapy is applied under the MR-linac. The breast surgery is planned after recovery from radiation induced acute toxicity, within 14 days. The surgeons would undertake lumpectomy only or an additional oncoplastic surgery, with axillary nodal evaluation with sentinal nodal biopsy or dissection. After wound healing, postoperative whole breast radiotherapy is administered, within 6 weeks following surgery. The dose is 26Gy/5.2Gy/5 fractions. Adjuvant systemic therapy is held until the end of the radiotherapy, no more than 12 weeks from surgery implementation.

ELIGIBILITY:
Inclusion Criteria:

1. Patients diagnosed with invasive breast cancer;
2. cN0 based on clinical physical examination combined with at least two imaging tests, or axillary fine-needle biopsy proved pN0;
3. Patients who plan to receive breast-conserving surgery or breast-conserving oncoplastic surgery;
4. No distant metastasis;
5. The primary tumour> 5mm from the skin, without invasion of the ribs or intercostal muscles;
6. No neoadjuvant systemic therapy;
7. Patients who can tolerate MRI;
8. Life expectancy ≥5 years;
9. Organ function is fine (Hemoglobin ≥100g/L, leukocyte ≥2×109/L, neutrophil ≥1×109/L, platelet ≥80×109/L; Creatinine 1.5 mg/dl or less; Alanine aminotransferase/aspartate aminotransferase ≤2.5×UNL.);
10. Patients are willing to cooperate to follow up;
11. Patients should sign the informed consent;
12. Women of childbearing age need effective contraception.

Exclusion Criteria:

1. Concurrent active connective tissue disease;
2. Patients who had radiotherapy to the ipsilateral breast or adjacent areas before;
3. Other malignancies, which affect pateint life expectancy (except adequately treated basal cell carcinoma of the skin, carcinoma in situ of the cervix, superficial bladder neoplasms (no more than T1));
4. Severe comorbidities or active disease (Poorly controlled heart disease: New York Classification of Cardiac Function ≥ Grade 2, active coronary heart disease, unstable angina pectoris, arrhythmia requiring medical treatment/persistent refractory hypertension; Myocardial infarction, stroke within six months; Poorly controlled diabetes persists. Fasting blood glucose ≥ 10mmol/L, 2 hours postprandial blood glucose ≥ 13 mmol/L. Poorly controlled psychosis develops or worsens within six months; Active infection; Positive for antibodies to HIV).

Max Age: 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 102 (Estimated)
Dates: Start 2022-06-21 (Actual); Primary Completion 2026-07-19 (Estimated); Study Completion 2028-07 (Estimated)

PRIMARY OUTCOMES:
The rate of patients who develop radiation-associated acute toxicity (≥ 2 degree) | until 4 weeks of postoperative radiotherapy
  We will record the incidence of ≥ 2 degree radiation-associated acute toxicity, such as breast or chest wall oedema, acute dermatitis, breast pain,itch of breast skin. The incidence of all the above is the primary outcome.

SECONDARY OUTCOMES:
Local recurrence rate | Until 5 years after diagnosis.
  The incidence of recurrence of any invasive or non-invasive breast cancer in the ipsilateral breast.
Local regional recurrence rate | Until 5 years after diagnosis.
  The incidence of recurrence in the ipsilateral breast or the lymphatic nodal regions.
Disease-free survival | Until 5 years after diagnosis.
  The time interval from diagnosis to any event of recurrence or death.
Overall survival | Until 5 years after diagnosis.
  The time interval from diagnosis to death from any reason.
Complications of surgery in the short term. | Until 30 days after the surgery.
  We will record the incidence of surgery assciated mobilidy events within 30 days, including bleeding, seroma, hematoma, wound dehiscence, flap necrosis, delayed wound healing, fat necrosis, wound infection, abscess and upper limb edema.
Quality of Life (according the outcomes of questionnaires to evaluate the quality of life) EORTC QLQ-C30 | Until 5 years after treatment.
  European Organization Research and Treatment of Cancer Breast Cancer-Specific Quality of Life Questionnaire EORTC QLQ-C30 to record patients' quality of life in different time points.
Quality of Life (according the outcomes of questionnaires to evaluate the quality of life) EORTC BR-23 | Until 5 years after treatment.
  European Organization for Research and Treatment of Cancer Breast Cancer-Specific Quality of Life Questionnaire EORTC BR-23 to record patients' quality of life in different time points.
Cosmetic outcome Breast Cancer Treatment Outcome Scale (BCTOS) | Until 5 years after treatment.
Cosmetic outcome Body Image Scale (BIS) | Until 5 years after treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Jing Wang, M.D., Study Chair — Cancer Institute and Hospital, Chinese Academy of Medical Sciences; Shu-lian Wang, M.D., Study Chair — Cancer Institute and Hospital, Chinese Academy of Medical Sciences; Hao Jing, M.D., Principal Investigator — Cancer Institute and Hospital, Chinese Academy of Medical Sciences; Xiang-yi Kong, M.D., Study Director — Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Locations (1):
- National Cancer Center/National Clinical Research Center for Cancer/Cancer Hospital, Chinese Academy of Medical Sciences and Peking Union Medical College, Beijing, Beijing Municipality, China

REFERENCES:
- [Derived] Dong H, Jing H, Wang XY, Kong XY, Wang YP, Zhai YR, Che SN, Fang Y, Wang SL, Wang J. Exploring the feasibility of preoperative tumor-bed boost, oncoplastic surgery, and adjuvant radiotherapy schedule in early-stage breast cancer: a phase II clinical trial. Int J Surg. 2025 Jan 1;111(1):382-393. doi: 10.1097/JS9.0000000000002073. PMID 39264581